CLINICAL TRIAL: NCT04419948
Title: Acute Effect of Oleocanthal Rich Extra-virgin Olive Oil on Postpranial Hyperglycemia and Platelet Activation of T2DM Patients
Brief Title: Oleocanthal Rich Olive Oil Acute Effects on Hyperglycemia and Platelet Activation in T2DM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harokopio University (Other)
Collaborators: National and Kapodistrian University of Athens (Other); University of Peloponnese (Other)
Responsible Party: Principal Investigator, Tzortzis Nomikos, Assistant Professor of Biochemistry, Harokopio University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 79549/16-05-2019
Record Dates: First submitted 2020-02-24; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Diabetes Mellitus, Adult-Onset; Platelet Dysfunction; Postprandial Hyperglycemia; Lipidemia; Inflammation; Oxidative Stress
Keywords: type 2 diabetes mellitus; diabetic platelet; platelet aggregation; oxidative stress; inflammation; postrpandial; hyperglycemia; extra virgin olive oil; oleocanthal; polyphenols; dyslipidemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia; Hyperlipidemias; Inflammation; Dyslipidemias | interventions — Butter; oleocanthal; Ibuprofen

STUDY DESIGN:
Intervention Model Description: Acute postprandial study with a randomized cross-over design
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (Experimental): 100g white bread plus 40ml butter
  Interventions: Other: White bread; Other: Butter
- Positive control (Experimental): 100g white bread plus 40ml butter and 400mg ibuprofen
  Interventions: Other: White bread; Other: Butter; Other: Ibuprofen
- Refined olive oil (Experimental): 100g white bread plus 40ml refined olive oil
  Interventions: Other: White bread; Other: Refined olive oil
- EVOO with moderate concentration of oleocanthal (Experimental): 100g white bread plus 40ml EVOO containing 250 mg/kg oleocanthal
  Interventions: Other: White bread; Other: EVOO with 250 mg/kg oleocanthal
- EVOO with high concentration of oleocanthal (Experimental): 100g white bread plus 40ml EVOO containing 500 mg/kg oleocanthal
  Interventions: Other: White bread; Other: EVOO with 500 mg/kg oleocanthal

INTERVENTIONS:
Other: White bread — White bread (120g) containing 54 g CHO
Other: Butter — Butter 39 g
  Arms: Control; Positive control
Other: Refined olive oil — Refined olive oil (40 ml).
  Arms: Refined olive oil
Other: EVOO with 250 mg/kg oleocanthal — Extra virgin olive oil containing 250 mg/kg oleocanthal.
  Arms: EVOO with moderate concentration of oleocanthal
Other: EVOO with 500 mg/kg oleocanthal — Extra virgin olive oil containing 500 mg/kg oleocanthal.
  Arms: EVOO with high concentration of oleocanthal
Other: Ibuprofen — Ibuprofen 400 mg
  Arms: Positive control

SUMMARY:
This is a pilot acute dietary intervention study with a randomized cross-over design aiming to investigate whether acute supplementation of extra virgin olive oil (EVOO) rich in oleocanthal could attenuate postprandial hyperglycemia and activation of platelets in T2DM patients. For this reason, non-insulin dependent diabetic patients (10-15) will be randomly assigned to consume in five different days white bread (50 g CHO) with butter, butter with ibuprofen, refined olive oil and olive oil with oleocanthal (250 mg/Kg 500 mg/Kg). Blood samples will be collected pre- and post-intervention up to 4 hours in order to determine platelet aggregation, postprnadial glycemia, lipemia, inflammation and oxidative stress.

Taking into account the strong anti-inflammatory and anti-platelet properties of oleocanthal, this study will assess whether oleocanthal-rich olive oils could exert similar effects under real in vivo conditions in T2DM patients. It will also assess whether these effects are achieved through improvement of postprandial glycemia and lipemia.

ELIGIBILITY:
Inclusion Criteria:

* adult patients diagnosed with T2DM
* stable weight the last two months
* smokers or not
* no restriction regarding the menopause

Exclusion Criteria:

* insulin therapy
* antiplatelet, anti-coagulant, anti-inflammatory and anti-depressant medication
* chronic inflammatory disease
* autoimmune diseases
* cancer
* uncontrolled thyroid disease.
* supplement consumption the last two months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-05-16 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of ADP-induced platelet aggregation at 90 min after meals consumption | 0 and 90 after the consumption of each type of meal
  EC50 (microM) of ADP induced platelet aggregation will be assessed by light transmittance aggregometry
Change from baseline of ADP-induced platelet aggregation at 240 min after meals consumption | 0 and 240 after the consumption of each type of meal
  EC50 (microM) of ADP induced platelet aggregation will be assessed by light transmittance aggregometry
Change from baseline of TRAP-induced platelet aggregation at 90 min after meals consumption | 0 and 90 after the consumption of each type of meal
  EC50 (microM) of TRAP induced platelet aggregation will be assessed by light transmittance aggregometry
Change from baseline of TRAP-induced platelet aggregation at 240 min after meals consumption | 0 and 240 after the consumption of each type of meal
  EC50 (microM) of TRAP induced platelet aggregation will be assessed by light transmittance aggregometry
Change from baseline of PAF-induced platelet aggregation at 90 min after meals consumption | 0 and 90 after the consumption of each type of meal
  EC50 (microM) of PAF induced platelet aggregation will be assessed by light transmittance aggregometry
Change from baseline of PAF-induced platelet aggregation at 240 min after meals consumption | 0 and 240 after the consumption of each type of meal
  EC50 (microM) of PAF induced platelet aggregation will be assessed by light transmittance aggregometry
Incremental Area Under the Serum Concentration Versus Time Curve (AUC) of Glucose | 0, 15, 30, 60, 90 120, 180, 240 min after the consumption of each meal
  iAUC of postprandial glucose will be calculated by serum glucose levels (mg/dL) which will be assessed by commercially available kits
Incremental Area Under the Serum Concentration Versus Time Curve (AUC) of Insulin | 0, 15, 30, 60, 90 120, 180, 240 min after the consumption of each meal
  iAUC of postprandial insulin will be calculated by serum insulin levels (mIU/L) which will be assessed by commercially available kits
Incremental Area Under the Serum Concentration Versus Time Curve (AUC) of Triglycerides | 0, 15, 30, 60, 90 120, 180, 240 min after the consumption of each meal
  iAUC of postprandial triglycerides will be calculated by serum triglyceride levels (mg/dL) which will be assessed by commercially available kits

SECONDARY OUTCOMES:
Incremental Area Under the Serum Concentration Versus Time Curve (AUC) of IL-6 | 0, 60, 120, 180, 240 min after the consumption of each meal
  iAUC of postprandial IL-6 will be calculated by serum IL-6 levels (mg/dL) which will be assessed by commercially available ELISA kits
Incremental Area Under the Plasma Concentration Versus Time Curve (AUC) of Protein Carbonyls | 0, 60, 120, 180, 240 min after the consumption of each meal
  iAUC of postprandial protein carbonyls will be calculated by plasma protein carbonyl levels (mg/dL) which will be determined by a photometric assay

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nutrition and Dietetics, Harokopio University, Athens, I Am Not in the U.S. Or Canada, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agrawal K, Melliou E, Li X, Pedersen TL, Wang SC, Magiatis P, Newman JW, Holt RR. Oleocanthal-rich extra virgin olive oil demonstrates acute anti-platelet effects in healthy men in a randomized trial. J Funct Foods. 2017 Sep;36:84-93. doi: 10.1016/j.jff.2017.06.046. Epub 2017 Jul 3. PMID 29904393